CLINICAL TRIAL: NCT05445947
Title: Enhancing And Supporting Early Development to Better Children's Lives (EASEL) Trial
Acronym: EASEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Nikolaos Sevdalis, Academic Director, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NUS-IRB-2021-993
Record Dates: First submitted 2022-06-24; First posted 2022-07-06 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Child Development
Keywords: educator; teacher; preschool; child; classroom

STUDY DESIGN:
Intervention Model Description: The EASEL trial will employ a Type 2 hybrid implementation-effectiveness design using a cluster randomized controlled trial. A hybrid design approach involves the simultaneous evaluation of both a programme's outcomes as well as the effectiveness of the implementation of the programme. A Type 2 hybrid design also enables the assessment of the feasibility of the programme. As part of the trial, 12 childcare centres will be randomized to receive training in the EASEL Approach (six sites, referred to as the intervention sites) or continue with business-as-usual (BAU) (six sites). Educators in the BAU group will be provided the option to be trained in the EASEL Approach following completion of the study.
Who Masked: Outcomes Assessor
Masking Description: The centers will be randomized by the research team to the intervention group (five to six centers) or control group (five to six centers) using a random number generator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Educators working at childcare centers in the intervention group will be trained and provided with ongoing coaching in the EASEL Approach.
  Interventions: Behavioral: The EASEL (Enhancing And Supporting Early Development to Better Children's Lives) Approach
- Control Group (No Intervention): Educators in the control group will continue with business-as-usual. Control group educators will be offered the opportunity to receive training in the EASEL Approach after completion of the trial.

INTERVENTIONS:
Behavioral: The EASEL (Enhancing And Supporting Early Development to Better Children's Lives) Approach — The EASEL Approach consists of a set of educator-led practices that can be incorporated into the daily classroom environment for children three to six years of age. The overall purpose of this approach is to enhance early childhood educators' teaching practices that would promote children's SEB+EF development.
  Nine EASEL practices were selected for inclusion in the EASEL Approach. These are a) core fundamental practices that are evidence-based, b) practices that expert stakeholders identified as ones for which local early childhood educators may need additional training, c) practices that are not already covered in pre-service training to avoid replication for educators, d) a combination of practices that educators may already be implementing and can enhance, and new practices, and e) a balance of antecedent and consequential practices (i.e., practices that can be implemented before and after a target behavior).
  Arms: Intervention Group

SUMMARY:
In The Lancet's series on advancing early childhood development, provision of high-quality early childhood care and education was listed as one of the main factors that can maximize children's potential to succeed in later life, particularly children from vulnerable or disadvantaged backgrounds. High-quality early childhood care and education is widely understood to be important for equipping children with essential skills and competencies across academic and non-academic areas, which in turn increases school readiness and has long-reaching impacts on outcomes later in life. Despite the government's efforts to support the early childhood sector, educators in Singapore continue to report difficulties in implementing practices in classrooms that promote children's social, emotional and cognitive development. To enhance educators' skills in these domains, we developed the Enhancing and Supporting Early development to better children's Lives (EASEL) Approach, a set of universal educator-led practices for use with 3-6-year-old children to improve social, emotional, behavioral and executive functioning (SEB+EF) outcomes. This study will evaluate the implementation and effectiveness of the EASEL Approach on improving early childhood educators' teaching practices and in turn, children's SEB+EF outcomes. We will conduct a type 2 hybrid implementation-effectiveness design in a cluster randomized controlled trial in 10-12 childcare centers. We will use the EPIS (Explore, Prepare, Implement, Sustain) Framework to support the implementation of the EASEL Approach. Implementation strategies include training, educator self-assessments, practice-based coaching, and data monitoring. Primary outcomes include educator's teaching practices and their adoption of the EASEL Approach in everyday practice. Secondary outcomes include the acceptability and feasibility of the EASEL Approach and children's SEB+EF outcomes. Quantitative and qualitative data will be collected at baseline, three months and six months.

DETAILED DESCRIPTION:
The specific aims of the EASEL trial are two-fold:

1. The first aim is to test the effectiveness of the EASEL Approach, a universal classroom-based approach (evidence-based classroom practices identified using a common elements approach) on enhancing educators' classroom practices to improve SEB+EF outcomes in preschool children. We hypothesize that the EASEL Approach will improve educators' teaching practices related to promoting preschool children's SEB+EF outcomes. In turn, improvements in children's outcomes in these domains in the longer term (e.g., six months) will also be observed.
2. The second aim of the trial is to understand how educators implement the EASEL Approach within their classroom and the factors that affect the implementation. We hypothesize that with the use of the implementation strategies proposed for the trial (educator training, educator self-assessment of intention to use and self-efficacy, practice-based coaching, and data monitoring), the EASEL Approach will be well adopted by educators, implemented sustainably and achieve its desired effects.

The EASEL trial is based on three key studies.

* The Growing Up in Singapore Towards healthy Outcomes (GUSTO) Study: A longitudinal birth cohort study of maternal and child health indicating significant relationships between conditions during pregnancy and early childhood on later outcomes of physical, mental and social well-being.
* McLeod et al. (2017): This trial builds on the systematic review to identify common elements considered for inclusion as part of the EASEL Approach.
* Work conducted by Assistant Professor Evelyn Law and colleagues at NUS Yong Loo Lin School of Medicine: The Whole Child Panel (WCP) 2.1 will be used in the EASEL trial as a screening measure of children's executive functioning and the Executive Function Playbook will be included as one of the EASEL practices.

The EASEL trial will employ a Type 2 hybrid implementation-effectiveness design using a cluster randomized controlled trial. A hybrid design approach involves the simultaneous evaluation of both a programme's outcomes as well as the effectiveness of the implementation of the programme. A Type 2 hybrid design also enables the assessment of the feasibility of the programme.

As part of the trial, 12 childcare centres will be randomized to receive training in the EASEL Approach (six sites, referred to as the intervention sites) or continue with business-as-usual (BAU) (six sites). Educators in the BAU group will be provided the option to be trained in the EASEL Approach following completion of the study.

The EASEL trial will be guided by the EPIS (Explore, Prepare, Implement, Sustain) Framework, an evidence-informed framework frequently used in programme implementation and evaluation. The EPIS Framework considers the multilevel nature of service systems (e.g., the early childhood sector in Singapore), the organizations within systems (e.g., individual preschool operators in Singapore), and the 'client' needs (e.g., the needs of children and early childhood educators) when implementing a new programme. It highlights four key phases that guide and describe the implementation process: Exploration, Preparation, Implementation, Sustainment. The Exploration phase involves identifying the problem, developing appropriate and evidence-based solutions, and considering factors that might impact implementation. In this context, the problem is the gap in educators' skills to enhance children's SEB+EF development, and the solution is the EASEL Approach. The Preparation phase consists of a planning process with key stakeholders (e.g., relevant government agencies, preschool operators, individual childcare centers) for the implementation of the new programme. When sufficient preparation has occurred, the Implementation phase commences (implementation of the EASEL Approach by educators in their classrooms). Factors affecting implementation include outer and inner contextual issues (e.g., resource availability, fit with educators' current practices, organizational culture, and attitudes) and consumer concerns (e.g., the applicability of practices for educators' and children's needs). When the new practices have been routinely used, the Sustainment phase can begin. This involves the sustainment of the new programme in the current setting and may also include scaling-up to other settings and systems.

ELIGIBILITY:
Inclusion Criteria:

For childcare centres:

* The childcare centre provides full-day programming for children at the Nursery 2 (N2), Kindergarten 1 (K1), and Kindergarten 2 (K2) levels (i.e., children between 3-5 years old at the start of the school year).Childcare centre has one of each class level that can participate in the EASEL trial (e.g., one N2, one K1 and one K2 class in each childcare centre).
* Childcare centre is not currently implementing other substantial SEB/EF programmes or involved in other trials evaluating SEB/EF programmes

For early childhood educators (adults):

* Both L1 and L2 educators will be eligible to take part in the trial. Inclusion of educators with a variety of experience will allow the research team to understand the effectiveness of various implementation strategies for each group. L1 educators are certified by the Early Childhood Development Agency (ECDA: government regulatory body for early childhood education) for deployment at nursery, pre-nursery and playgroup (i.e., children aged 18 months-4 years old) and L2 educators are certified by ECDA for deployment at kindergarten, nursery, pre-nursery and playgroup (i.e., children aged 18 months-6 years old).
* Educators must be ECDA-certified English-language educators.

For children:

* Children must be enrolled in N2, K1 or K2 classes at the start of the trial.
* Child is attending the participating childcare centre, in the selected class.
* Child is enrolled to attend a full-day childcare programme.

For parents/caregivers:

* Parent/caregiver needs to be the primary caregiver of the target child in the study.
* Parent/caregiver needs to be able to read/write in English. Where parents/caregivers are not proficient in English, their consent will be sought with the aid of interpreters, but data will only be collected for their child via teacher reports.

Exclusion Criteria:

For childcare centres:

* Childcare centre does not have at least 1 class at each age level (N2, K1 and K2 level).
* Childcare centre is currently implementing other substantial SEB/EF programmes or involved in other trials evaluating SEB/EF programmes.
* Childcare centre is currently involved in other research trials.
* Childcare centre currently has areas of concerns flagged to ECDA for review.

For early childhood educators (adults):

* Educator does not have either L1 or L2 certification
* Educator does not teach primarily in English.

For children:

* Child attends only a half-day or flexi childcare programme.

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Change in educator's teaching practices and classroom quality | Pre-intervention (i.e., baseline - before training workshop), post-intervention (i.e., 6-month)
  The Early Childhood Classroom Observation Measure (ECCOM; Stipek & Byler, 2004) is an observational assessment that involves a 3-hour classroom observation by a trained researcher. Domains on the ECCOM include Management, Climate, and Classroom Instruction. Subdomains under Management include Child Responsibility, Classroom Management, Choices of Activities and Discipline Strategies; subdomains under Climate include Support for Communication Skills, Support for Interpersonal Skills, Student Engagement, Individualization of Learning Activities, and Educator Warmth/Responsiveness; subdomains under Instruction include Learning Standards, Coherence of Instructional Activities, Teaching Concepts, Instructional Conversation and Relevance of Activities to Children's Experience.
Change in children's social-emotional development, behaviour and self-regulation skills | Pre-intervention (i.e., baseline), post-intervention (i.e., 6-month)
  The Child Self-Regulation and Behavior Questionnaire (CSBQ; Howard & Melhuish, 2017) is a 34-item self-report questionnaire for educators to indicate the option that best fits what each child is like (1 = Not True to 5 = Very True). Items on the CSBQ cover the following domains: Self-regulation (cognitive, emotional, behavioral), Sociability, Prosocial Behavior, Externalizing and Internalizing Behavior, and General Child Development.
Change in children's executive functioning | Pre-intervention (i.e., baseline), post-intervention (i.e., 6-month)
  The Behavior Rating Inventory of Executive Functioning - Preschool version (BRIEF-P; Gioia et al., 2003) is a 63-item self-report questionnaire for parents to indicate how often a child has had problems with various behaviors in the past six months (0 = Never, 1 = Sometimes, 2 = Often). The BRIEF-P consists of the following indices: Inhibitory Self-Control Index, Flexibility Index, Emergent Metacognition Index, and Global Executive Composite; and the following domains: Inhibit, Shift, Emotional Control, Working Memory, Plan/Organize.
Children's executive functioning (screening) | Post-intervention (i.e., 6-month)
  The executive functioning tasks from the Singapore Whole Child Panel 2.1 (WCP 2.1) will be administered by the research team with the child to measure executive functioning skills such as working memory and cognitive flexibility. These tasks will take about 10 minutes and will be administered using an electronic device: '8 Boxes' and 'Day and Night'. The WCP 2.1 is a screening measure which will only be administered at the post-intervention timepoint.
Change in educator's uptake of EASEL Approach (Intervention Group only) | Pre-intervention (i.e., baseline - after training workshop), mid-intervention (i.e., 3-month), post-intervention (i.e., 6-month)
  Educator self-assessments will be used to assess educators' (1) attitudes toward the EASEL practices, (2) perceived norms of the EASEL practices, (3) intentions to use the EASEL practices, and (4) self-efficacy with the EASEL practices.
Frequency and educator's uptake of online EASEL resources (Intervention Group only) | Post-intervention (i.e., 6-month)
  Frequency and uptake of online EASEL resources will be assessed through educators' engagement data on Thinkific (e.g., number of times lessons were accessed and completed).
Educator's uptake and adoption of EASEL Approach (Intervention Group only) | Post-intervention (i.e., 6-month)
  Focus group discussions with groups of key stakeholders (i.e., center leadership and educators in the Intervention Group)

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Sevdalis, PhD, Principal Investigator — NUS Singapore
Locations (4):
- Singapore (4):
  - M.Y. World, Singapore
  - PAP Community Foundation, Singapore
  - Presbyterian Preschool Services, Singapore
  - Skool4Kidz, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] The Lancet. Advancing early childhood development: From science to scale: An executive summary for The Lancet's series. Lancet. 2016;389(10064):1-8.
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] McLeod BD, Sutherland KS, Martinez RG, Conroy MA, Snyder PA, Southam-Gerow MA. Identifying Common Practice Elements to Improve Social, Emotional, and Behavioral Outcomes of Young Children in Early Childhood Classrooms. Prev Sci. 2017 Feb;18(2):204-213. doi: 10.1007/s11121-016-0703-y. PMID 27562037
- [Background] Aarons GA, Hurlburt M, Horwitz SM. Advancing a conceptual model of evidence-based practice implementation in public service sectors. Adm Policy Ment Health. 2011 Jan;38(1):4-23. doi: 10.1007/s10488-010-0327-7. PMID 21197565
- [Background] Fishman J, Beidas R, Reisinger E, Mandell DS. The Utility of Measuring Intentions to Use Best Practices: A Longitudinal Study Among Teachers Supporting Students With Autism. J Sch Health. 2018 May;88(5):388-395. doi: 10.1111/josh.12618. PMID 29609213
- [Background] Fishman J, Lushin V, Mandell DS. Predicting implementation: comparing validated measures of intention and assessing the role of motivation when designing behavioral interventions. Implement Sci Commun. 2020 Sep 28;1:81. doi: 10.1186/s43058-020-00050-4. eCollection 2020. PMID 33005900
- [Background] Maddox BB, Crabbe SR, Fishman JM, Beidas RS, Brookman-Frazee L, Miller JS, Nicolaidis C, Mandell DS. Factors Influencing the Use of Cognitive-Behavioral Therapy with Autistic Adults: A Survey of Community Mental Health Clinicians. J Autism Dev Disord. 2019 Nov;49(11):4421-4428. doi: 10.1007/s10803-019-04156-0. PMID 31385175
- [Background] Pellecchia M, Beidas RS, Marcus SC, Fishman J, Kimberly JR, Cannuscio CC, Reisinger EM, Rump K, Mandell DS. Study protocol: implementation of a computer-assisted intervention for autism in schools: a hybrid type II cluster randomized effectiveness-implementation trial. Implement Sci. 2016 Nov 25;11(1):154. doi: 10.1186/s13012-016-0513-4. PMID 27884169
- [Background] Stipek D, Byler P. The early childhood classroom observation measure. Early Child Res Q. 2004;19(3):375-97.
- [Background] Law EC, Chong SC, Nadarajan R, Broekman BFP, Rifkin-Graboi A, Shorey S, et al. Pediatrics and the multidimensional nature of school readiness: A population-based study.
- [Background] Vasarri S, Isquith PK. Development of the Behavior Rating Inventory of Executive Function - Preschool Version (Brief-P) in 10 Languages. Value Health. 2014 Nov;17(7):A575. doi: 10.1016/j.jval.2014.08.1933. Epub 2014 Oct 26. No abstract available. PMID 27201927
- [Background] Howard SJ, Melhuish E. An Early Years Toolbox for Assessing Early Executive Function, Language, Self-Regulation, and Social Development: Validity, Reliability, and Preliminary Norms. J Psychoeduc Assess. 2017 Jun;35(3):255-275. doi: 10.1177/0734282916633009. Epub 2016 Feb 28. PMID 28503022
- [Background] Bierman KL, Torres M. Promoting the development of executive functions through early education and prevention programs. In: Executive function in preschool-age children: Integrating measurement, neurodevelopment, and translational research. 2015. p. 299-326.
- [Background] O'Connor EE, Dearing E, Collins BA. Teacher-child relationship and behavior problem trajectories in elementary school. Am Educ Res J [Internet]. 2011 Feb 1 [cited 2021 Feb 10];48(1):120-62. Available from: http://journals.sagepub.com/doi/10.3102/0002831210365008
- [Background] Carter AS, Briggs-Gowan MJ, Davis NO. Assessment of young children's social-emotional development and psychopathology: recent advances and recommendations for practice. J Child Psychol Psychiatry. 2004 Jan;45(1):109-34. doi: 10.1046/j.0021-9630.2003.00316.x. PMID 14959805
- [Background] Diamond A. Executive functions. Annu Rev Psychol. 2013;64:135-68. doi: 10.1146/annurev-psych-113011-143750. Epub 2012 Sep 27. PMID 23020641
- [Background] McCain MN, Mustard JF, Shanker S. Early Years Study 2: Putting science into action. Toronto, Canada; 2007.
- [Background] Ang L, Lipponen L, May Yin SL. Critical reflections of early childhood care and education in Singapore to build an inclusive society. Policy Futur Educ [Internet]. 2020 Nov 23 [cited 2020 Dec 7];147821032097110. Available from: http://journals.sagepub.com/doi/10.1177/1478210320971103
- [Background] Lipponen L, Lim S. Vital voices for vital years. 2019.
- [Background] Bautista A, Ng SC, Múñez D, Bull R. Learning areas for holistic education: kindergarten teachers' curriculum priorities, professional development needs, and beliefs. Int J Child Care Educ Policy [Internet]. 2016 Dec 1 [cited 2021 Jan 5];10(1):8. Available from: https://ijccep.springeropen.com/articles/10.1186/s40723-016-0024-4
- [Background] Taylor MJ, McNicholas C, Nicolay C, Darzi A, Bell D, Reed JE. Systematic review of the application of the plan-do-study-act method to improve quality in healthcare. BMJ Qual Saf. 2014 Apr;23(4):290-8. doi: 10.1136/bmjqs-2013-001862. Epub 2013 Sep 11. PMID 24025320
- [Derived] Tan ES, McLeod BD, Mildon RA, Shlonsky A, Seah CKF, McCrickerd K, Goh E, Kembhavi G. Assessing the effectiveness and implementation of a universal classroom-based set of educator practices to improve preschool children's social-emotional outcomes: Protocol for a cluster randomized controlled type 2 hybrid trial in Singapore. PLoS One. 2023 Sep 20;18(9):e0291723. doi: 10.1371/journal.pone.0291723. eCollection 2023. PMID 37729260

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT05445947/Prot_SAP_000.pdf